CLINICAL TRIAL: NCT06844825
Title: The Effectiveness of Telerehabilitation Versus In-Person Rehabilitation in Managing Chronic Low Back Pain: a Pragmatic Randomized Non-Inferiority Trial
Brief Title: Telerehabilitation in Managing Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shibili Nuhmani, Assistant Porfessor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-PGS-2025-03-0019
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain (LBP)
MeSH Terms: conditions — Low Back Pain | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele rehabilitation (Experimental)
  Interventions: Other: Tele rehabilitation
- Usual care (Active Comparator)
  Interventions: Other: usual care only

INTERVENTIONS:
Other: Tele rehabilitation — The experimental group will receive the treatment remotely by ZOOM platform and phone call
  Arms: Tele rehabilitation
Other: usual care only — in-person usual care provided by the physical therapist
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether telerehabilitation is as effective as in-person rehabilitation in treating patients with chronic back pain in actual clinical practice settings.T he study will recruit eighty-four individuals with chronic LBP, who will be randomly assigned to one of two groups: telerehabilitation (TR) or the control group, who will receive standard clinic therapy. The TR group will be treated remotely via phone calls and the Zoom platform. The intervention program will be customized according to the requirements and abilities of each patient. It will include self-management skills, education and support, including Pain Neuroscience Education , and customized exercises.

ELIGIBILITY:
Inclusion Criteria: Adults aged 18 and above with non-specific chronic low back pain more than 12 weeks.

Exclusion Criteria: Cancer, systematic or neurological diseases, fracture, recent surgery on the spine and/or extremities, cognitive impairment, pregnant women, and communication barriers or other medical conditions contraindicating TR. If there is any presence of red flags, such as cauda equina syndrome, spinal infection, spinal compression fractures, spinal stress fractures, ankylosing spondylitis, or aneurysm will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain | baseline and immediately after the intervention
  Pain measured by numeric rating scale
function | baseline and immediately after the intervention
  measured by the Oswestry function index

IPD SHARING:
Plan to Share IPD: Undecided